CLINICAL TRIAL: NCT04998500
Title: Growth Hormone as a Model for Reversible Activation of Adipose Tissue Fibrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aarhus (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1-10-72-283-20
Record Dates: First submitted 2021-08-09; First posted 2021-08-10 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Fibrosis
Keywords: Adipose tissue; Fibrosis; Growth hormone; Fibro-adipogenic progenitors
MeSH Terms: conditions — Fibrosis | interventions — Growth Hormone; Sodium Chloride; pegvisomant

STUDY DESIGN:
Intervention Model Description: This study aims to uncover physiological in vivo effects of growth hormone (GH). The intervention with GH and Pegvisomant will therefore be used as tools to activate a well-known physiological response.
  Participants are randomized to receive either control intervention first and then GH intervention, or GH intervention first and then control intervention.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GH intervention - control intervention (Experimental): Participants will receive daily subcutaneous injections of growth hormone for 7 days. Approximately 1-4 months later, the participants will receive daily subcutaneous injections of control intervention for 7 days consisting of saline and GH receptor blockade (Pegvisomant).
  Interventions: Biological: Growth hormone, saline and GH receptor blockade (Pegvisomant)
- Control intervention - GH intervention (Experimental): Participants will receive daily subcutaneous injections of control intervention for 7 days consisting of saline and GH receptor blockade (Pegvisomant). Approximately 1-4 months later, the participants will receive daily subcutaneous injections of growth hormone for 7 days.
  Interventions: Biological: Growth hormone, saline and GH receptor blockade (Pegvisomant)

INTERVENTIONS:
Biological: Growth hormone, saline and GH receptor blockade (Pegvisomant) — This study aims to uncover physiological effects of growth hormone (GH). The intervention with GH and GH receptor blockade (Pegvisomant) will therefore be used as tools to activate a well-known physiological response. Thus, this study is not a drug trial.

SUMMARY:
Background: Adipose tissue fibrosis denotes excessive pathological accumulation of extracellular matrix (ECM) in adipose tissue and is a marker of dysfunction. Growth hormone (GH) activates adipose tissue lipolysis and stimulates collagen synthesis in lean tissues. Intriguingly, we have novel pilot data to suggest that GH excess (acromegaly) also induces reversible fibrosis in vivo and potently activates the expression of fibroblast activation protein alpha (FAPα).

Hypothesis: GH induces adipose tissue fibrosis by increased FAPα expression together with proliferation and fibrogenic differentiation of fibro-adipogenic progenitor (FAP) cells.

Aim: To unravel the mechanisms underlying GH-induced adipose tissue fibrosis with emphasis on FAPα expression and proliferation of FAP cells.

Subjects and methods: In a single blinded, randomized, double-dummy crossover design, 10 adult, moderately overweight individuals will be subjected to one week of GH and GH receptor blockade (Pegvisomant). We will use single-cell technologies, fluorescence-activated cell sorting (FACS), RNA sequencing, and cell culture studies on adipose tissue samples, combined with in vivo assessment of adipose tissue turnover and metabolism.

Perspectives: Understanding fibrosis formation in human models may identify new targets for treatment of obesity-associated disorders.

DETAILED DESCRIPTION:
Background and preliminary data: Adipose tissue is a multicellular tissue surrounded by an extracellular matrix, which undergoes continuous remodeling. Pertubations in the remodeling processes may cause accumulation of excess extracellular matrix protein and hence fibrosis. Adipose tissue fibrosis is recognized as a component of the metabolic syndrome together with insulin resistance, dyslipidemia and obesity, and fibrosis is likely to play a causative role (1,2). In this context, it is fascinating that prolonged GH exposure in vivo induces insulin resistance despite a concomitant mobilization and reduction of fat mass (3). This effect of GH is expressed in patients with a GH-producing pituitary tumor (acromegaly) (4). Moreover, GH is a potent activator of collagen turnover and it also promotes fibrosis in human tendons and skeletal muscles (5-7). Increased AT fibrosis has been reported in a GH transgenic mice model (8) and we have preliminary data showing AT fibrosis in patients with active acromegaly, which reverses after disease control.

Little is known about the mechanisms underlying GH-induced fibrosis, but recent evidence points to a potential involvement of FAPα, an enzyme that is highly expressed in mouse AT FAP cells (9). Moreover, we have recently reported that human skeletal muscle FAP cells upregulate FAPα (DPP4) during fibrogenic differentiation (19). FAPα is a subunit of a heterodimeric proteinase complex attached to the cell membrane in addition to a soluble form also present in the circulation (10). Several proteins are recognized as FAPα substrates, including collagen type I (11) and III (12), and FAPα appears to play a significant role in hepatic tissue remodeling (13) and in lung fibrosis (14). We have recently recorded elevated circulating levels of FAPα in active acromegaly, which correlates with collagen turnover reverses after disease control (15). Fibro-adipogenic progenitor cells are mesenchymal progenitors with the intrinsic potential to differentiate into either collagen-producing fibroblasts or adipocytes. They have been studied in murine cardiac and skeletal muscle, where they contribute to either fibrosis or fat deposition during muscle-impaired regeneration or degeneration (16-18). We have recently demonstrated that a subset of FAP cells drives the accumulation of ECM protein and adipocytes in the muscle from patients with type 2 diabetes and likely contributes to the poor metabolic and mechanical muscle function (19). Whether GH affects adipose tissue FAP cell proliferation and differentiation is unknown, but FAP cell proliferation is regulated by IGF-I (16), which is a strongly GH-dependent peptide. Increased FAP proliferation has also been reported to contribute to intramuscular adipose tissue (IMAT) in several conditions, and we have observed IMAT after treatment in acromegaly (unpublished data). Furthermore, we have preliminary data from FACS-isolated adipose tissue FAP cells incubated with serum from acromegaly patients, which suggest GH-dependent increased FAP cell proliferation and fibrogenic appearance. Collectively, these findings suggest that GH promotes a pro-proliferative and fibrogenic FAP phenotype at the expense of adipogenic differentiation.

Hypotheses: Growth hormone: 1) Activates FAPα protein expression, 2) Increases proliferation and fibrogenic differentiation of FAP cells, and 3) Induces reversible fibrosis in adipose tissue in humans

Subjects and methods: In a single blinded, randomized, double-dummy crossover design, 10 adult, moderately overweight individuals will be subjected to one week of GH and GH receptor blockade (Pegvisomant). Pegvisomant is a modfied GH molecule that selectively blocks the GH receptor and is a licensed drug for the treatment of acromegaly. We include Pegvisomant as an 'active control' in order to suppress endogenous GH actions. The participants will receive daily subcutaneous injections of growth hormone, 0.6-2.0 mg depending on age, for 7 days in the GH intervention. In the control intervention, the participants will receive daily subcutaneous injections of either Pegvisomant or saline. Pegvisomant in a dose of 30 mg is given two times, in the beginning and in the end of the control intervention, whereas saline is given on the other 5 days of the control intervention period. The two intervention periods are separated by a wash out period of 1-4 months. The participants will be randomized to either start with the GH intervention and next be subjected to the control intervention, or start with the control intervention and next be subjected to the GH intervention. The participants will meet at the hospital daily for the injections and a small blood sample. Each intervention period is initiated by an initiation day where there will be taken blood samples, adipose tissue and muscle samples, be performed temperature measurements and bioimpedance, and be administered heavy water and the first injection of intervention either GH or control intervention. On the first initiation day a DXA scan will be performed for assessment of body composition. Each intervention period will be terminated with a study day where there will be taken blood samples, adipose tissue and muscle samples, be performed temperature measurements, indirect calorimetry, palmitate tracer kinetics and bioimpedance, and be administered the last injection of intervention either GH or control intervention. The participants will be fasting for the initiation and study days, and during the intervention periods, they will log their intake of food and beverages.

Study outcomes:

Primary: FAP cell function, FAPα protein expression and markers of fibrosis in AT biopsies obtained before and after intervention. In particular, we will perform:

* FACS to quantify and isolate cell populations, including quantification of FAP cells in adipose tissue, and in vitro determination of proliferation and fibro-/adipogenic differentiation potential
* FAPα expression in blood and adipose tissue
* Markers of fibrosis in adipose tissue assessed by light microscopy and immunohistochemically, RNA sequencing and heavy water labeled connective tissue turnover

Secondary: to study the impact of GH exposure on:

* Circulating biomarkers of collagen turnover (PINP, PIIINP)
* Whole body energy metabolism and fatty acid turnover (indirect calorimetry and palmitate tracer kinetics)
* Connective tissue turnover in muscle tissue (heavy water (D2O) labeling)
* Temperature measurements

Statistical analysis plan: Comparison between groups will be performed using standard statistical methods (t-test or equivalent nonparametric test). Within group comparison will be performed using paired t-test of equivalent nonparametric test. Moreover, ANOVA (repeated measures) will be used. A p-value less than 0.05 will be regarded as statistically significant.

Perspective and relevance: This is the first study to investigate GH effects on adipose tissue fibrosis in humans, which has implications beyond GH pathophysiology. A deeper understanding of the pathways controlling fibroblast and adipocyte balance in fat tissue is essential groundwork and may unravel new targets for combating adipose tissue dysfunction and related disorders. As recently demonstrated in type 2 diabetic patients these progenitor cells are key mediators of tissue plasticity and function in humans (19).

ELIGIBILITY:
Inclusion Criteria:

* Written and oral consent before enrollment
* Legally competent subjects
* Healthy (except uncomplicated hypertension and hypercholesterolemia)
* Male sex
* Age ≥ 18 years and ≤ 50 years
* BMI 25-35

Exclusion Criteria:

* Any condition which the investigator considers might affect the participant's ability to complete the study
* Known of presumed acute of chronic illness

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Fibro-adipogenic progenitor (FAP) cells | Anticipated approximately 1-5 months
  Quantification of FAP cells in adipose tissue, and in vitro determination of proliferation and fibro-/adipogenic differentiation potential
Fibroblast activation protein (FAPα) | Anticipated approximately 1-5 months
  FAPα concentration and activity in blood, and expression in adipose tissue
Adipose tissue fibrosis | Anticipated approximately 1-5 months
  Markers of fibrosis in adipose tissue assessed by light microscopy and immunohistochemically, RNA sequencing and heavy water labeled connective tissue turnover

SECONDARY OUTCOMES:
Circulating biomarkers of collagen turnover | Anticipated approximately 1-5 months
  (PINP, PIIINP)
Protein turnover in muscle tissue | Anticipated approximately 1-5 months
  Heavy water labeled protein and connective tissue turnover in muscle tissue to compare with protein turnover in adipose tissue
Metabolism and fatty acid turnover | Anticipated approximately 1-5 months
  Whole body energy metabolism and fatty acid turnover (indirect calorimetry and palmitate tracer kinetics)
Temperature | Anticipated approximately 1-5 months
  Temperature measurements

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Bæk, MD, Principal Investigator — University of Aarhus; Jens Otto L Jørgensen, Professor, Study Director — University of Aarhus
Locations (1):
- Aarhus University, Aarhus, Denmark

REFERENCES:
- [Background] Munoz A, Abate N, Chandalia M. Adipose tissue collagen and inflammation in nonobese Asian Indian men. J Clin Endocrinol Metab. 2013 Aug;98(8):E1360-3. doi: 10.1210/jc.2012-3841. Epub 2013 Jun 18. PMID 23780376
- [Background] Lawler HM, Underkofler CM, Kern PA, Erickson C, Bredbeck B, Rasouli N. Adipose Tissue Hypoxia, Inflammation, and Fibrosis in Obese Insulin-Sensitive and Obese Insulin-Resistant Subjects. J Clin Endocrinol Metab. 2016 Apr;101(4):1422-8. doi: 10.1210/jc.2015-4125. Epub 2016 Feb 12. PMID 26871994
- [Background] Moller N, Jorgensen JO. Effects of growth hormone on glucose, lipid, and protein metabolism in human subjects. Endocr Rev. 2009 Apr;30(2):152-77. doi: 10.1210/er.2008-0027. Epub 2009 Feb 24. PMID 19240267
- [Background] Melmed S. Acromegaly pathogenesis and treatment. J Clin Invest. 2009 Nov;119(11):3189-202. doi: 10.1172/JCI39375. Epub 2009 Nov 2. PMID 19884662
- [Background] Longobardi S, Keay N, Ehrnborg C, Cittadini A, Rosen T, Dall R, Boroujerdi MA, Bassett EE, Healy ML, Pentecost C, Wallace JD, Powrie J, Jorgensen JO, Sacca L. Growth hormone (GH) effects on bone and collagen turnover in healthy adults and its potential as a marker of GH abuse in sports: a double blind, placebo-controlled study. The GH-2000 Study Group. J Clin Endocrinol Metab. 2000 Apr;85(4):1505-12. doi: 10.1210/jcem.85.4.6551. PMID 10770189
- [Background] Doessing S, Heinemeier KM, Holm L, Mackey AL, Schjerling P, Rennie M, Smith K, Reitelseder S, Kappelgaard AM, Rasmussen MH, Flyvbjerg A, Kjaer M. Growth hormone stimulates the collagen synthesis in human tendon and skeletal muscle without affecting myofibrillar protein synthesis. J Physiol. 2010 Jan 15;588(Pt 2):341-51. doi: 10.1113/jphysiol.2009.179325. Epub 2009 Nov 23. PMID 19933753
- [Background] Doessing S, Holm L, Heinemeier KM, Feldt-Rasmussen U, Schjerling P, Qvortrup K, Larsen JO, Nielsen RH, Flyvbjerg A, Kjaer M. GH and IGF1 levels are positively associated with musculotendinous collagen expression: experiments in acromegalic and GH deficiency patients. Eur J Endocrinol. 2010 Dec;163(6):853-62. doi: 10.1530/EJE-10-0818. Epub 2010 Sep 21. PMID 20858702
- [Background] Householder LA, Comisford R, Duran-Ortiz S, Lee K, Troike K, Wilson C, Jara A, Harberson M, List EO, Kopchick JJ, Berryman DE. Increased fibrosis: A novel means by which GH influences white adipose tissue function. Growth Horm IGF Res. 2018 Apr;39:45-53. doi: 10.1016/j.ghir.2017.12.010. Epub 2017 Dec 20. PMID 29279183
- [Background] Merrick D, Sakers A, Irgebay Z, Okada C, Calvert C, Morley MP, Percec I, Seale P. Identification of a mesenchymal progenitor cell hierarchy in adipose tissue. Science. 2019 Apr 26;364(6438):eaav2501. doi: 10.1126/science.aav2501. PMID 31023895
- [Background] Hamson EJ, Keane FM, Tholen S, Schilling O, Gorrell MD. Understanding fibroblast activation protein (FAP): substrates, activities, expression and targeting for cancer therapy. Proteomics Clin Appl. 2014 Jun;8(5-6):454-63. doi: 10.1002/prca.201300095. Epub 2014 Mar 24. PMID 24470260
- [Background] Park JE, Lenter MC, Zimmermann RN, Garin-Chesa P, Old LJ, Rettig WJ. Fibroblast activation protein, a dual specificity serine protease expressed in reactive human tumor stromal fibroblasts. J Biol Chem. 1999 Dec 17;274(51):36505-12. doi: 10.1074/jbc.274.51.36505. PMID 10593948
- [Background] Christiansen VJ, Jackson KW, Lee KN, McKee PA. Effect of fibroblast activation protein and alpha2-antiplasmin cleaving enzyme on collagen types I, III, and IV. Arch Biochem Biophys. 2007 Jan 15;457(2):177-86. doi: 10.1016/j.abb.2006.11.006. Epub 2006 Nov 17. PMID 17174263
- [Background] Levy MT, McCaughan GW, Marinos G, Gorrell MD. Intrahepatic expression of the hepatic stellate cell marker fibroblast activation protein correlates with the degree of fibrosis in hepatitis C virus infection. Liver. 2002 Apr;22(2):93-101. doi: 10.1034/j.1600-0676.2002.01503.x. PMID 12028401
- [Background] Fan MH, Zhu Q, Li HH, Ra HJ, Majumdar S, Gulick DL, Jerome JA, Madsen DH, Christofidou-Solomidou M, Speicher DW, Bachovchin WW, Feghali-Bostwick C, Pure E. Fibroblast Activation Protein (FAP) Accelerates Collagen Degradation and Clearance from Lungs in Mice. J Biol Chem. 2016 Apr 8;291(15):8070-89. doi: 10.1074/jbc.M115.701433. Epub 2015 Dec 9. PMID 26663085
- [Background] Arlien-Soborg MC, Grondahl C, Baek A, Dal J, Madsen M, Hogild ML, Pedersen SB, Bjerre M, Jorgensen JOL. Fibroblast Activation Protein is a GH Target: A Prospective Study of Patients with Acromegaly Before and After Treatment. J Clin Endocrinol Metab. 2020 Jan 1;105(1):dgz033. doi: 10.1210/clinem/dgz033. PMID 31544947
- [Background] Farup J, Madaro L, Puri PL, Mikkelsen UR. Interactions between muscle stem cells, mesenchymal-derived cells and immune cells in muscle homeostasis, regeneration and disease. Cell Death Dis. 2015 Jul 23;6(7):e1830. doi: 10.1038/cddis.2015.198. PMID 26203859
- [Background] Joe AW, Yi L, Natarajan A, Le Grand F, So L, Wang J, Rudnicki MA, Rossi FM. Muscle injury activates resident fibro/adipogenic progenitors that facilitate myogenesis. Nat Cell Biol. 2010 Feb;12(2):153-63. doi: 10.1038/ncb2015. Epub 2010 Jan 17. PMID 20081841
- [Background] Uezumi A, Fukada S, Yamamoto N, Takeda S, Tsuchida K. Mesenchymal progenitors distinct from satellite cells contribute to ectopic fat cell formation in skeletal muscle. Nat Cell Biol. 2010 Feb;12(2):143-52. doi: 10.1038/ncb2014. Epub 2010 Jan 17. PMID 20081842
- See also: Reference number 19 — https://pubmed.ncbi.nlm.nih.gov/34678202/